CLINICAL TRIAL: NCT07318389
Title: ASCEND-CRC: Profiling and Targeting Dynamic Tumor Resistance in Patients With Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1634; NCI-2025-09705 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-12-30; First posted 2026-01-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Dynamic Tumor Resistance; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Standard of Care; Bevacizumab; Cetuximab; Panitumumab; IFL protocol; Folfox protocol; encorafenib; adagrasib; Trifluridine; tipiracil; trifluridine tipiracil drug combination; trastuzumab deruxtecan; tucatinib; sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASCEND-CRC Sample Collection (Experimental): Standard of care
  Interventions: Other: SOC (Standard of care); Drug: Bevacizumab; Drug: Cetuximab; Drug: Panitumumab; Drug: FOLFIRI; Drug: FOLFOX; Drug: Encorafenib; Drug: Adagrasib; Drug: Trifluridine/tipiracil (TAS-102); Drug: Trastuzumab deruxtecan; Drug: Tucatinib; Drug: Sotorasib

INTERVENTIONS:
Other: SOC (Standard of care) — Blood draws, biopsies, samples and MRI.
Drug: Bevacizumab — Given by IV
Drug: Cetuximab — Given by Iv
Drug: Panitumumab — Given by Iv
Drug: FOLFIRI — Given by Iv
Drug: FOLFOX — Given by Iv
Drug: Encorafenib — Given by po
Drug: Adagrasib — Given by Po
Drug: Trifluridine/tipiracil (TAS-102) — Given by po
Drug: Trastuzumab deruxtecan — Given by IV
Drug: Tucatinib — Given by po
Drug: Sotorasib — Given by po

SUMMARY:
To find out if certain drug/therapy combinations that are targeted to individual patients based on characteristics of their disease types may help to control the disease.

DETAILED DESCRIPTION:
Primary Objectives

* To determine differences in PFS based on differential response markers in paired tissue biopsies (Part I).
* To improve progression-free survival with novel intervention strategies (Part II)

Secondary Objectives

* To collect serial tissue and blood biomarkers and efficacy data associated with standard of care or investigational therapy across multiple lines of therapy.
* To determine the overall response rate (ORR), and overall survival (OS) based on the presence of specific biomarkers or adaptive interventions.

ELIGIBILITY:
Eligibility Criteria

* The participant has a histologically or cytologically confirmed diagnosis of colorectal cancer.
* Confirmation of non-MSI-H/pMMR status.
* Tumor that is measurable as per RECIST v1.1 and biopsy able, defined as lesion/tumor that can be biopsied without undue risk.
* Age ≥ 18 years.
* ECOG performance status 0-2.
* Due to the potential teratogenic effect of chemotherapy, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for an adequate amount of time following end of treatment based on the SOC indications for the administered regimen (Refer to Pregnancy Assessment Policy MD Anderson Institutional

Policy # CLN1114). This includes all female participants, between the onset of menses and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

  * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for an adequate amount of time following end of treatment based on the SOC indications for the administered regimen.
  * The participant is willing and able to sign the informed consent in compliance with protocol requirements, including mandatory biopsies.

Exclusion Criteria

* Pregnancy.
* Participants with concurrent or recent (less than 1 year before consent) malignancies that have the potential to interfere with the study safety and/or endpoint assessments will be excluded.
* Participants for whom there is an intent to proceed to curative therapy (i.e., resection) will be excluded.
* Participants who have undergone treatment with both oxaliplatin and irinotecan in the metastatic setting will be excluded. Treatment with oxaliplatin in the adjuvant setting with relapse within 6 months will be counted as treatment in the metastatic setting for the purpose of this criterium.
* For participants who have undergone treatment for metastatic disease, participants who have not progressed (clinically or radiographically) on the most recent therapy will be excluded.
* Concurrent participation in any other interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-06-10 (Estimated); Primary Completion 2027-11-14 (Estimated); Study Completion 2029-11-14 (Estimated)

PRIMARY OUTCOMES:
safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org